CLINICAL TRIAL: NCT02336399
Title: Sustained HBsAg and Viral Response in Patients Achieved HBsAg Loss by Interferon Treatment
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Yao Xie, Liver Diseases Center, Beijing Ditan Hospital
Other Study IDs: DTXY002
Record Dates: First submitted 2015-01-08; First posted 2015-01-13 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Chronic Hepatitis B
Keywords: HBsAg loss, interferon, HBV reaction
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for HBV serological and HBV DNA testing
Oversight: Data Monitoring Committee: No

SUMMARY:
Chronic hepatitis B (CHB) is a serious liver disease worldwide, and the leading cause of cirrhosis and hepatocellular carcinoma (HCC).HBsAg loss/seroconversion is considered to be the ideal endpoint of antiviral therapy in both HBeAg-positive and HBeAg-negative patients, as well as the ultimate treatment goal in CHB. However, some patients who have achieved HBsAg loss would reverse back to HBsAg positive, or even become HBV reactive with recurrence of viremia. In current study, the viral and HBsAg response in patients who have achieved HBsAg loss by interferon (IFN) treatment will be observed for 96 weeks after the completion of IFN treatment. The primary analysis will be performed at the end of 96 weeks. Following the completion of the study period of 96 weeks, patients will be offered to participate in a long term study for further observation of additional 144 weeks (total of 240 weeks from the enrollment).

DETAILED DESCRIPTION:
Chronic hepatitis B patients who have achieved HBsAg loss from interferon treatment will be enrolled and observed for 96 weeks. Serum HBV DNA, HBsAg, anti-HBs, HBeAg, and anti-HBe will be measured every 3 months during the observation period. Their liver function and chemistry tests are also performed every 3 months. The liver ultrasonic examination would be taken every 3-6 months. The primary measurement is the percentage of patients who have positive HBsAg and/or a detectable level of HBV DNA. Following the completion of the study period, patients will be offered to participate in a long term study for further observation of additional 144 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had chronic hepatitis B and achieved HBsAg loss by interferon treatment.

Exclusion Criteria:

* Active consumption of alcohol and/or drugs
* Co-infection with human immunodeficiency virus, hepatitis C virus, or hepatitis D virus
* History of autoimmune hepatitis
* Psychiatric disease
* Evidence of neoplastic diseases of the liver

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population in this study is composed of patients who have chronic hepatitis B and achieved HBsAg loss from interferon treatment. Eligible patients will have serum HBsAg and HBV DNA tests every 3 months for 96 weeks after finishing the interferon treatment. The sustained HBsAg response is defined as the levels of serum HBsAg mantaining below the low level of quantitation and the levels of HBV DNA remain undetectable. Following the completion of the study period, patients will be offered to participate in a long term study for further observation up to 240 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 420 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
The rate of sustained HBsAg negativity and viral response in 96 weeks | From the enrollment to 96 weeks
  The percentage of patients who have both undetectable level of HBsAg and undetectable level of serum HBV DNA at 96 weeks after completing treatment with interferon

SECONDARY OUTCOMES:
The rate of sustained HBsAg negativity and viral response in long term | From the enrollment to 240 weeks
  The percentage of patients who have both undetectable level of HBsAg and undetectable level of serum HBV DNA at 240 weeks after completing treatment with interferon
The rate of sustained HBsAg negativity and viral response in subset analysis in 96 weeks | From the enrollment to 96 weeks
  The percentage of patients who have both undetectable level of HBsAg and undetectable level of serum HBV DNA at 96 weeks after completing treatment with interferon mono-therapy versus those who have the same endpoints after the completion of the interferon therapy in the combination or sequencing of oral antiviral therapy
The rate of sustained HBsAg negativity and viral response in subset analysis for long term | From the enrollment to 240 weeks
  The percentage of patients who have both undetectable level of HBsAg and undetectable level of serum HBV DNA at 240 weeks after completing treatment with interferon mono-therapy versus those who have the same endpoints after completing the interferon therapy in the combination or sequencing of oral antiviral therapy
Predictor(s) for recurrence of HBsAg positivity or detectable levels of HBV DNA in 96 weeks | From the enrollment to 96 weeks
  Clinical features and baseline factors will be analyzed by comparing patients who have sustained HBsAg negativity and viral response vs. those who have no sustained endpoints at week 96.
Predictor(s) for recurrence of HBsAg positivity or detectable levels of HBV DNA in long term | From the enrollment to 240 weeks
  Clinical features and baseline factors will be analyzed by comparing patients who have sustained HBsAg negativity and viral response vs. those who have no sustained endpoints at week 240.

OTHER OUTCOMES:
Exploratory outcomes on complication rates of liver cancer and decompensated cirrhosis in 96 weeks | from the enrollment to the 96 weeks
  Percentage of patient who have clinical cirrhosis or liver cancer during the observational period
Exploratory outcomes on complication rates of liver cancer and decompensated cirrhosis in 240 weeks | from the enrollment to the 240 weeks
  Percentage of patient who have clinical cirrhosis or liver cancer during the observational period

CONTACTS AND LOCATIONS:
Overall Officials: Yao Xie, MD, Principal Investigator — Beijing Ditan Hospital, Beijing, China
Locations (1):
- Beijing Ditan Hospital,Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Pan CQ, Li MH, Yi W, Zhang L, Lu Y, Hao HX, Wan G, Cao WH, Wang XY, Ran CP, Shen G, Wu SL, Chang M, Gao YJ, Xie Y. Outcome of Chinese patients with hepatitis B at 96 weeks after functional cure with IFN versus combination regimens. Liver Int. 2021 Jul;41(7):1498-1508. doi: 10.1111/liv.14801. Epub 2021 Feb 16. PMID 33486874